CLINICAL TRIAL: NCT01018823
Title: A Phase 1, Randomized, Placebo-Controlled, Parallel Group, 14 Day Repeated Dose Escalation Study To Evaluate The Safety, Tolerability, Pharmacokinetics, And Pharmacodynamics Of PF-04971729 In Otherwise Healthy Overweight And Obese Adult Subjects
Brief Title: A Multiple Dose Study Of Ertugliflozin (PF-04971729, MK-8835) In Otherwise Healthy Overweight And Obese Volunteers (MK-8835-037)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 8835-037
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — ertugliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Ertugliflozin 1 mg (Experimental): Ertugliflozin 1 mg, oral, once daily for 14 days
  Interventions: Drug: Ertugliflozin
- Ertugliflozin up to 5 mg (Experimental): Ertugliflozin up to 5 mg, oral, once daily for 14 days
  Interventions: Drug: Ertugliflozin
- Ertugliflozin up to 25 mg (Experimental): Ertugliflozin up to 25 mg, oral, once daily for 14 days
  Interventions: Drug: Ertugliflozin
- Ertugliflozin up to 100 mg (Experimental): Ertugliflozin up to 100 mg, once daily for 14 days
  Interventions: Drug: Ertugliflozin
- Placebo (Placebo Comparator): Placebo to Ertugliflozin once daily for 14 days
  Interventions: Drug: Placebo to Ertugliflozin

INTERVENTIONS:
Drug: Ertugliflozin — Ertugliflozin oral dosing 1 mg, 5 mg, 25 mg, or 100 mg solutions/suspensions administered once daily for 14 days immediately after breakfast
  Other Names: PF-04971729; MK-8835
  Arms: Ertugliflozin 1 mg; Ertugliflozin up to 100 mg; Ertugliflozin up to 25 mg; Ertugliflozin up to 5 mg
Drug: Placebo to Ertugliflozin — Placebo oral dosing solutions/suspensions administered once daily for 14 days immediately after breakfast
  Arms: Placebo

SUMMARY:
Ertugliflozin (PF-04971729, MK-8835) is under development for the treatment of Type 2 Diabetes. The primary purpose of this trial is to evaluate the safety and tolerability, pharmacokinetics and pharmacodynamics, of multiple oral doses of ertugliflozin.

DETAILED DESCRIPTION:
To evaluate the safety and tolerability, pharmacokinetics (PK), and pharmacodynamics, of multiple oral doses of ertugliflozin.

ELIGIBILITY:
Inclusion Criteria:

Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive.

Body Mass Index (BMI) of 26.5 to 35.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).

Evidence of glycosuria, as defined by a positive urine dipstick test; Fasting (at least 10 hours) serum triglyceride >300 mg/dL; Fasting (at least 10 hours) LDL-cholesterol >190 mg/dL; Fasting (at least 10 hours) serum 25-OH Vitamin D concentration <20 ng/mL

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2009-12-14 (Actual); Primary Completion 2010-03-18 (Actual); Study Completion 2010-03-18 (Actual)

PRIMARY OUTCOMES:
Number of Participants Experiencing an Adverse Event (AE) | Up to 28 days postdose (Up to 42 days)
Number of Participants Discontinuing Study Drug Due to an AE | Up to 14 days
Area under the plasma concentration-time curve (AUC) over the dosing interval tau (AUCtau) for ertugliflozin | Up to 17 days
Maximum plasma concentration (Cmax) of ertugliflozin | Up to 17 days
Time taken to reach the maximum observed plasma concentration (Tmax) of ertugliflozin | Up to 17 days
Ertugliflozin half life (t1/2) | Up to 17 Days
Apparent clearance (CL/F) after a single dose of ertugliflozin | Up to 17 days
Apparent volume of distribution (Vz/F) | Up to 17 days
Observed Accumulation Ratio of Area Under the Curve for the dosing interval of ertugliflozin (Rac[obs]) | Up to 17 days
Change from baseline in 24-hour weighted mean glucose | Baseline and Day 14
Change from baseline in 24-hour urinary glucose excretion | Baseline and Day 14
Change from baseline in 24-hour plasma C-peptide | Baseline and Day 14
Inhibition of glucose reabsorption | Baseline and Day 14
Change from baseline in body weight | Baseline and Day 14
Area under the plasma concentration-time curve over 8 hours (AUC[0-8]) for serum intact parathyroid hormone | Up to 17 days
Area under the plasma concentration-time curve over 24 hours (AUC[0-24]) for serum intact parathyroid hormone | Up to 17 days
Trough concentration of serum intact parathyroid hormone (Ctrough) | Up to 17 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Fediuk DJ, Nucci G, Dawra VK, Cutler DL, Amin NB, Terra SG, Boyd RA, Krishna R, Sahasrabudhe V. Overview of the Clinical Pharmacology of Ertugliflozin, a Novel Sodium-Glucose Cotransporter 2 (SGLT2) Inhibitor. Clin Pharmacokinet. 2020 Aug;59(8):949-965. doi: 10.1007/s40262-020-00875-1. PMID 32337660
- [Derived] Marshall JC, Liang Y, Sahasrabudhe V, Tensfeldt T, Fediuk DJ, Zhou S, Krishna R, Dawra VK, Wood LS, Sweeney K. Meta-Analysis of Noncompartmental Pharmacokinetic Parameters of Ertugliflozin to Evaluate Dose Proportionality and UGT1A9 Polymorphism Effect on Exposure. J Clin Pharmacol. 2021 Sep;61(9):1220-1231. doi: 10.1002/jcph.1866. Epub 2021 Jun 19. PMID 33813736